CLINICAL TRIAL: NCT04507607
Title: Efficacy and Safety of TAF in Pregnant Women With Chronic Hepatitis B Infection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chaoshuang Lin, Professor Lin, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0237801
Record Dates: First submitted 2020-07-18; First posted 2020-08-11 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Chronic Hepatitis B; Mother-to-child Block; Antiviral Treatment
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women with CHB (Experimental): Start taking TAF at 24 weeks of gestation until delivery. The liver function, viral load and antigen status were reviewed monthly and 10 ml peripheral blood was collected.
  Interventions: Drug: Tenofovir Alafenamide 25 MG
- women with CHB (Active Comparator): Nonpregnant women taking TAF for antiviral therapy were regularly rechecked for liver function, viral load, and antigens.
  Interventions: Drug: Tenofovir Alafenamide 25 MG

INTERVENTIONS:
Drug: Tenofovir Alafenamide 25 MG — TAF was administered to pregnant women with CHB during pregnancy for mother-to-child interention.Women with chronic hepatitis B who are not pregnant receive TAF for antiviral treatment.

SUMMARY:
The effectiveness of mother-to-child block of CHB in pregnant women in the middle and later stages of pregnancy has been recognized by the guidelines. TAF, as a newly marketed antiviral drug, has not been conclusively concluded in terms of its efficacy and postpartum safety in preventing mother-to-child transmission in pregnant women.Our purpose is to explore the TAF for CHB the curative effect of pregnant and postnatal security.

DETAILED DESCRIPTION:
After diagnosis at the infection clinic of the Third Affiliated Hospital of Sun Yat-sen University, the eligible patients were enrolled into the group.Each person will sign the informed consent prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* 25 pregnant women with HBeAg (+), HBV DNA ≥ 2*10^6IU/mL who met the diagnostic criteria in the guidelines for the prevention and treatment of chronic hepatitis B were pregnant women at 24-28 weeks of pregnancy.
* 25 non-pregnant women with HBeAg (+), HBV DNA ≥ 2*10^6IU/mL who met the diagnostic criteria in the guidelines for the prevention and treatment of chronic hepatitis B.
* The enrolled patients were all newly admitted patients without treatment, and if they did not meet the standard after completing the relevant examination, they would be removed.

Exclusion Criteria:

* Coinfection with HAV, HCV, HDV, HEV or HIV;
* A history of antiviral therapy or concurrent treatment with immunoregulatory drugs, antitumor drugs, cytotoxic drugs or immunosuppressive steroids;
* Three-dimensional ultrasonography showed fetal malformation;
* The spouse is infected with HBV;
* History of decompensated liver disease (e.g., decompensated liver disease with coagulation disorders, hyperbilirubinemia, hepatic encephalopathy, hypoalbuminemia, ascites and esophageal varicose bleeding), history of liver cancer or other chronic liver disease (e.g., autoimmune hepatitis) or clinical symptoms;
* History of immune diseases;
* A history of serious cardiovascular disease;
* Other reasons the researchers considered it inappropriate to participate in the trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Liver indicators of intrapartum | intrapartum
  The level of liver function (ALT、AST)、HBV DNA、HBV Serological markers (HBsAg、HBeAg、HBeAb) in pregnant women at birth.
Liver indicators of postpartum | 12 months postpartum
  The level of liver function (ALT、AST)、HBV DNA、HBV Serological markers (HBsAg、HBeAg、HBeAb) in pregnant women 1 month、3 month、7 month、9 month、12 month after delivery.

SECONDARY OUTCOMES:
Liver indicators of pregnancy | 24 weeks gestation until delivery
  The level of liver function (ALT、AST)、HBV DNA、HBV Serological markers (HBsAg、HBeAg、HBeAb) in pregnant women taking TAF 0、4、8、12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- LinChaoshuang, Guangzhou, China